CLINICAL TRIAL: NCT04424238
Title: Clinical Research on Mobile Medical Used for the Standardized Management of Gestational Diabetes: a Randomized Control Trail
Brief Title: the Effect of Mobile Medical Used for the Standardized Management of Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JS-1012
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-05

CONDITIONS: GDM; Blood Glucose; Compliance, Patient; Diet Habit
Keywords: GDM; CGM; m-health; diet modification; blood glucose; compliance
MeSH Terms: conditions — Patient Compliance; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Clinic Prenatal Care (Control Group) (No Intervention): pregnancy's prenatal care appointment would be changed to once every two weeks when diagnosed with GDM. Doctors generally ask GDM women record their daily diet, exercise, weight, BG and blood pressure for at least three days between two visits and give lifestyle guidance according to the records. If they fail to show diaries, doctors would ask them come back with record next week. If BG control is poor, medicine intervention would be considered.
- m-health group (Intervention Group) (Experimental): participants were managed continuously through WeChat group chat.
  Interventions: Behavioral: m-health management

INTERVENTIONS:
Behavioral: m-health management — Patients in intervention group received additional WeChat group management when conducted standard clinic prenatal care.
  Arms: m-health group (Intervention Group)

SUMMARY:
A multicenter, randomized controlled trial was conducted to investigate whether health education and life style management through WeChat group chat was more effective in controlling blood glucose (BG) than standard clinic prenatal care in women with GDM.

DETAILED DESCRIPTION:
Most gestational diabetes mellitus (GDM) can be well controlled by health education and life style management, expecting a better pregnancy outcome. But standard clinic prenatal care which consist of clinic visit every two weeks may not give full play to the effects of GDM management. Telemedicine shows its potential to fill this gap. A multicenter, randomized controlled trial was designed to investigate whether health education and life style management through WeChat group chat was more effective in controlling blood glucose (BG) than standard clinic prenatal care in women with GDM. Women with GDM diagnosed by oral glucose tolerance test between 23-30+6 gestational weeks were randomized to a WeChat group chat-based blood glucose management group or routine clinic prenatal care. In PUMCH, investigators also equip CGM for m-health group allowing a more detailed BG information. The primary outcome was change of glycemic qualification rate during follow up period in both groups. The second outcome was pregnancy outcomes. Also, a case-control study is designed to compare the glucose control status between rice-richen meal and wheaten-richen meal, and all other macronutrients and micronutrients are all calculated and same between two groups, which may provide more clues for type of carbohydrate recommendation for Chinese women with GDM.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 45 years.
* With singleton pregnancy
* Diagnosed as GDM by 75g oral glucose tolerance test (OGTT) and insulin treatment is not required assessed by multi-disciplinary consultation.
* Be able to use smart phone for chatting, read and write basic Chinese.
* Volunteer for research.

Exclusion Criteria:

* Pregnancies with diagnosed chronic disease
* Pregnancies with other pregnancy complications except GDM
* Pregnancies had recent trauma and treatment of glucocorticoids

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
glycemic qualification rate | From enrollment to 42 days postpartum
  Glycemic qualification rate was calculated by the number of BG within the control range /30*100%. BG control range were fasting BG (fasting and before-sleep BG)<95 mg/dL (5.3 mmol/L) and two-hour postprandial BG (post-breakfast, post-lunch, post-dinner BG)<120 mg/dL (6.7 mmol/L)

SECONDARY OUTCOMES:
pregnancy outcome | delivery
  delivery mode, premature rupture of the membranes, preterm birth, birthweight and postpartum hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Liangkun Ma, Study Chair — Chinese Academy of Medical Science & Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No